CLINICAL TRIAL: NCT00034983
Title: A Worldwide, Multicenter, Double-Blind, Parallel, Active-Controlled, Long-Term Safety Study of MK0869 in Outpatients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-066)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-066; Formally-497B; MK0869-066; 2006_407
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: aprepitant
  Other Names: MK0869
Drug: Comparator: paroxetine HCL

SUMMARY:
A clinical study to determine the efficacy and safety of an investigational medication (MK0869) in the treatment of depression

DETAILED DESCRIPTION:
The duration of treatment is 1 year.

ELIGIBILITY:
Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2001-10-29 (Actual); Primary Completion 2003-12-29 (Actual); Study Completion 2003-12-29 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability. | Duration of treatment

SECONDARY OUTCOMES:
Sexual dysfunction adverse experiences and gastrointestinal disturbance adverse experiences | Duration of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Snyder E, Cai B, DeMuro C, Morrison MF, Ball W. A New Single-Item Sleep Quality Scale: Results of Psychometric Evaluation in Patients With Chronic Primary Insomnia and Depression. J Clin Sleep Med. 2018 Nov 15;14(11):1849-1857. doi: 10.5664/jcsm.7478. PMID 30373688